CLINICAL TRIAL: NCT07179692
Title: Clinical Study of CEA-Targeted Chimeric Antigen Receptor T Lymphocytes (CAR-T) in Advanced CEA-Positive Malignant Solid Tumors
Brief Title: CEA-Targeted CAR-T Therapy in CEA-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC094
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Gastric Cancer; Colon Cancer; Rectal Cancer; Esophageal Cancer; Pancreas Cancer
MeSH Terms: conditions — Lung Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-15x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells
- Intrapleural infusion of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-15x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells
- Intraperitoneal infusion of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 1-15x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T cells

INTERVENTIONS:
Biological: CEA-targeted CAR-T cells — Administration method: intravenous infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intravenous of CEA-targeted CAR-T
Biological: CEA-targeted CAR-T cells — Administration method: intrapleural infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intrapleural infusion of CEA-targeted CAR-T
Biological: CEA-targeted CAR-T cells — Administration method: intraperitoneal infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.
  Arms: Intraperitoneal infusion of CEA-targeted CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalating + dose-expansion clinical study, aiming to evaluate the safety and efficacy of CEA-targeted CAR-T cell preparations, and to preliminarily observe the study drug in CEA-positive advanced malignant tumors. The pharmacokinetic characteristics of CAR-T cell preparations for the treatment of patients with CEA-positive advanced malignancies were obtained and the recommended dose and infusion schedule.

DETAILED DESCRIPTION:
According to the different infusion methods, patients will be assigned to three parallel subgroups: intravenous infusion, intrapleural infusion, and intraperitoneal infusion.

Within each subgroup, the study is conducted in two sequential parts:

1. .Part A (dose-escalation): escalation begins at the lowest dose level; 3-6 subjects are enrolled at each dose level;
2. .Part B (dose-expansion): additional subjects are treated at the recommended dose identified in Part A to further evaluate safety and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restriction;
2. Histopathologically confirmed diagnosis of advanced, metastatic, or recurrent malignant tumors, primarily including colorectal cancer, esophageal cancer, gastric cancer, pancreatic cancer, lung cancer, and cholangiocarcinoma;
3. Failure of at least second-line standard treatment (disease progression or intolerance, such as surgery, chemotherapy, radiotherapy, etc.) or lack of effective treatment options;
4. Immunohistochemical staining of tumor samples showing CEA positivity (clear membrane staining, positivity rate ≥ 10%) within the past 3 months; if the immunohistochemical result is older than 3 months (clear membrane staining, positivity rate ≥ 10%), serum CEA must exceed 10 µg/L;
5. At least one evaluable lesion according to RECIST 1.1 criteria;
6. ECOG performance status of 0-2;
7. Expected survival of ≥ 12 weeks;
8. No severe psychiatric disorders;
9. Unless otherwise specified, the following important organ function criteria must be met:

   1. Hematology: White blood cells > 2.0 × 10^9/L, neutrophils > 0.8 × 10^9/L, lymphocytes > 0.5 × 10^9/L, platelets > 50 × 10^9/L, hemoglobin > 90 g/L;
   2. Cardiac function: Echocardiogram shows ejection fraction ≥ 50%, ECG shows no significant abnormalities;
   3. Renal function: Serum creatinine ≤ 2.0 × ULN;
   4. Liver function: ALT and AST ≤ 3.0 × ULN (can be relaxed to ≤ 5.0 × ULN for patients with liver tumor infiltration);
   5. Total bilirubin ≤ 2.0 × ULN;
   6. Oxygen saturation > 92% without supplemental oxygen;
10. Eligible for single or venous blood collection, and no contraindications for cell collection;
11. The subject agrees to use reliable and effective contraception methods from the time of signing the informed consent form until 1 year after CAR-T cell infusion (excluding rhythm method);
12. The subject or their authorized guardian agrees to participate in this clinical trial and signs the informed consent form (ICF), indicating understanding of the trial's purpose and procedures and willingness to participate in the study.

Exclusion Criteria:

1. Clinically symptomatic central nervous system metastasis or meningeal metastasis at screening, or other evidence indicating that central nervous system or meningeal metastasis has not been controlled, as determined by the investigator, making the patient unsuitable for enrollment.
2. Participation in another clinical trial within 1 month prior to screening.
3. Receipt of live attenuated vaccines within 4 weeks prior to screening.
4. Received the following anti-tumor treatments within 14 days or at least 5 half-lives (whichever is shorter) prior to screening: chemotherapy, targeted therapy, or other experimental drug treatments.
5. Active infection requiring systemic treatment or an uncontrolled infection.
6. Bowel obstruction, active gastrointestinal bleeding, or a history of major gastrointestinal bleeding within the last 3 months, or severe gastrointestinal conditions such as severe gastric or duodenal ulcers, severe ulcerative colitis, or other severe gastrointestinal inflammations.
7. Toxicity from prior anti-tumor treatments has not improved to baseline levels or ≤ grade 1, except for alopecia or peripheral neuropathy.
8. Any of the following cardiac conditions:

   1. New York Heart Association (NYHA) Class III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to enrollment;
   3. Clinically significant ventricular arrhythmias, or history of unexplained syncope (excluding cases due to vasovagal or dehydration);
   4. Severe non-ischemic cardiomyopathy.
9. Active autoimmune diseases or other conditions requiring long-term use of immunosuppressive therapy.
10. History of another malignancy within the past 3 years, excluding treated and stable in situ cervical cancer or basal cell carcinoma of the skin.
11. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA levels above the normal range; positive for hepatitis C virus (HCV) antibodies with peripheral blood HCV RNA levels above the normal range; positive for HIV antibodies; or positive for syphilis testing.
12. Pregnant or breastfeeding women.
13. Any other conditions that, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cell preparations in the treatment of CEA-positive advanced malignancies [Safety and Tolerability] | 1 month
  Incidence of adverse events during the study, evaluated per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) criteria
Obtained the recommended dose and infusion regimen of CAR-T cells for the treatment of patients with CEA-positive advanced malignancies[Safety and Tolerability] | 1 month
  Dose-limiting toxicity after CEA CAR-T cell infusion

SECONDARY OUTCOMES:
Assessing disease control rates of CAR-T cell preparations in CEA-positive advanced malignancies [Effectiveness] | From infusion through Month 3
  Disease control rate: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
To evaluate the efficacy of CAR-T cell preparations in CEA-positive advanced malignancies【Effectiveness】 | From infusion through Month 3
  Changes in serum tumor marker levels: CEA, CA19-9, CA-125, etc.
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  Cmax: maximum observed level of circulating CAR-T cells in peripheral blood after infusion
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  To determine the time to maximum observed level of circulating CAR-T cells (Tmax)
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  To estimate AUC0-28d and AUC0-90d for circulating CAR-T cells

OTHER OUTCOMES:
Objective response rate (ORR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Donglai Lv, MD, Principal Investigator — The 901 Hospital of Joint Logistics Support Force of People Liberation Army
Locations (1):
- The 901 Hospital of Joint Logistics Support Force of People Liberation Army, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No